CLINICAL TRIAL: NCT03931941
Title: A Phase 3 Open-Label Clinical Study to Evaluate the Safety and Tolerability of Rebiotix RBX2660 (Microbiota Suspension) in Subjects With Recurrent Clostridium Difficile Infection
Brief Title: Microbiota Restoration Therapy for Recurrent Clostridium Difficile Infection (PUNCH CD3-OLS)
Acronym: CD3-OLS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rebiotix Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-01
Record Dates: First submitted 2019-04-26; First posted 2019-04-30 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2023-04

CONDITIONS: Clostridium Difficile Infection; Infection; Communicable Diseases
Keywords: C. Difficile Diarrhea; Clostridium Difficile; CDI; FMT; Fecal Microbiota Transplant; Microbiota Restoration Therapy; Diarrhea; Microbial Suspension; Fecal Transplant; C Difficile Colitis; Clostridium Difficile Associated Diarrhea; C diff diarrhea; C Difficile; C diff
MeSH Terms: conditions — Clostridium Infections; Infections; Communicable Diseases; Diarrhea; Enterocolitis, Pseudomembranous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active (Experimental): RBX2660 is an enema of a microbiota suspension
  Interventions: Drug: RBX2660

INTERVENTIONS:
Drug: RBX2660 — RBX2660 is a microbiota suspension administered as an enema
  Other Names: Microbiota suspension

SUMMARY:
This is a prospective, multicenter, open-label Phase 3 study of a microbiota suspension of intestinal microbes. Patients who have had at least one recurrence of CDI after a primary episode and have completed at least one round of standard-of-care oral antibiotic therapy or have had at least two episodes of severe CDI resulting in hospitalization may be eligible for the study. Subjects may receive a second RBX2660 enema if they are deemed treatment failures following the initial enema per the protocol-specified treatment failure definition.

DETAILED DESCRIPTION:
This is a prospective, multicenter, open-label Phase 3 study of a microbiota suspension of intestinal microbes. The primary assessments for this study are (i) safety via assessment of treatment-emergent adverse events and (ii) efficacy of RBX2660 preventing recurrent episodes of CDI measured at 8 weeks after treatment. Follow-up office visits occur at 1 week and 8 weeks after completing the initial study treatment. Telephone assessments occur at 4 weeks, and 4 and 6 months after the study. Patients who have had at least one recurrence of CDI after a primary episode and have completed at least one round of standard-of-care oral antibiotic therapy or have had at least two episodes of severe CDI resulting in hospitalization may be eligible for the study. Subjects may receive a second RBX2660 enema if they are deemed treatment failures following the initial enema per the protocol-specified treatment failure definition.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old.
2. Medical record documentation of either: a) a current diagnosis or history of recurrent CDI as determined by the treating physician, b) or has had at least two episodes of severe CDI resulting in hospitalization.
3. Is currently taking or was just prescribed antibiotics to control CDI related diarrhea at the time of enrollment. [Note: Subject's CDI diarrhea must be controlled (<3 unformed/loose stools/day) while taking antibiotics during screening.]

Exclusion Criteria:

1. Has continued CDI diarrhea despite being on a course of antibiotics prescribed for CDI treatment.
2. Requires systemic antibiotic therapy for a condition other than CDI.
3. Fecal microbiota transplant (FMT) within the past 6 months.
4. FMT with an associated serious adverse event related to the FMT product or procedure.
5. Bezlotoxumab (CDI monoclonal antibodies) if received within the last year.
6. CD4 count <200/mm^3 during Screening.
7. An absolute neutrophil count of <1000 cells/µL during Screening.
8. Pregnant, breastfeeding, or intends to become pregnant during study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 793 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teena Chopra, M.D., M.P.H., Study Chair — Wayne State University
Locations (51):
- United States (46):
  - Phoenix, Phoenix, Arizona
  - North Little Rock, North Little Rock, Arkansas
  - Oxnard, Oxnard, California
  - Aurora, Aurora, Colorado
  - Hamden, Hamden, Connecticut
  - Gainesville, Gainesville, Florida
  - Jacksonville, Jacksonville, Florida
  - Naples, Naples, Florida
  - Orlando, Orlando, Florida
  - Port Orange, Port Orange, Florida
  - Atlanta, Atlanta, Georgia
  - Decatur, Decatur, Georgia
  - Idaho Falls, Idaho Falls, Idaho
  - Burr Ridge, Burr Ridge, Illinois
  - Gurnee, Gurnee, Illinois
  - Fort Wayne, Fort Wayne, Indiana
  - Wichita, Wichita, Kansas
  - New Orleans, New Orleans, Louisiana
  - Shreveport, Shreveport, Louisiana
  - Baltimore, Baltimore, Maryland
  - Detroit, Detroit, Michigan
  - Plymouth, Plymouth, Minnesota
  - Rochester, Rochester, Minnesota
  - St. Louis, St Louis, Missouri
  - New York, New York, New York
  - Rochester, Rochester, New York
  - Durham, Durham, North Carolina
  - Fargo, Fargo, North Dakota
  - Cleveland, Cleveland, Ohio
  - Oklahoma City, Oklahoma City, Oklahoma
  - Philadelphia, Philadelphia, Pennsylvania
  - Pittsburgh, Pittsburgh, Pennsylvania
  - Wyomissing, Wyomissing, Pennsylvania
  - Charleston, Charleston, South Carolina
  - Hixon, Hixon, Tennessee
  - Nashville, Nashville, Tennessee
  - Dallas, Dallas, Texas
  - Houston, Houston, Texas
  - West Jordan, West Jordan, Utah
  - Annandale, Annandale, Virginia
  - Springfield, Springfield, Virginia
  - Seattle, Seattle, Washington
  - Spokane, Spokane, Washington
  - Madison, Madison, Wisconsin
  - Marshfield, Marshfield, Wisconsin
  - Milwaukee, Milwaukee, Wisconsin
- Canada (5):
  - Calgary, Calgary, Alberta
  - Edmonton, Edmonton, Alberta
  - Vancouver, Vancouver, British Columbia
  - Victoria, Victoria, British Columbia
  - Moncton, Moncton, New Brunswick

REFERENCES:
- [Derived] Skinner AM, Lodise TP, Reilly J, Guthmueller B, Srivastava S, Axelrad JE. Safety and Efficacy of Fecal Microbiota, Live-jslm for Prevention of Recurrent Clostridioides difficile Infection Among Hospitalized Participants in PUNCH CD3-OLS. Infect Dis Ther. 2026 Feb 7. doi: 10.1007/s40121-026-01304-9. Online ahead of print. PMID 41653256
- [Derived] Lee C, Feuerstadt P, Louie T, Bancke L, Guthmueller B, Harvey A, Hoeyer F, Orenstein R, Dubberke ER, Khanna S. Integrated analysis of the safety of fecal microbiota, live-jslm in adults with recurrent Clostridioides difficile infection from five prospective clinical trials: an update. Therap Adv Gastroenterol. 2025 Nov 12;18:17562848251395566. doi: 10.1177/17562848251395566. eCollection 2025. PMID 41245385
- [Derived] Aroniadis OC, Guthmueller B, Dehlin K, Srivastava S, Feuerstadt P, Lembo A, Weber HC. Safety and Efficacy of Fecal Microbiota, Live-jslm to Prevent Recurrent Clostridioides difficile Infection in Participants With Irritable Bowel Syndrome. Infect Dis Ther. 2025 Sep;14(9):2157-2169. doi: 10.1007/s40121-025-01208-0. Epub 2025 Aug 10. PMID 40784972
- [Derived] Alonso CD, Tillotson GS, Bidell MR, Guthmueller B, Hoeyer F, Fischer M, Dubberke ER. Safety and Efficacy of Fecal Microbiota, Live-jslm, in Preventing Recurrent Clostridioides difficile Infection in Participants Who Were Mildly to Moderately Immunocompromised in the Phase 3 PUNCH CD3-OLS Study. Open Forum Infect Dis. 2025 Mar 4;12(4):ofaf117. doi: 10.1093/ofid/ofaf117. eCollection 2025 Apr. PMID 40177588
- [Derived] Feuerstadt P, Chopra T, Knapple W, Van Hise NW, Dubberke ER, Baggott B, Guthmueller B, Bancke L, Gamborg M, Steiner TS, Van Handel D, Khanna S. PUNCH CD3-OLS: A Phase 3 Prospective Observational Cohort Study to Evaluate the Safety and Efficacy of Fecal Microbiota, Live-jslm (REBYOTA) in Adults With Recurrent Clostridioides difficile Infection. Clin Infect Dis. 2025 Feb 5;80(1):43-51. doi: 10.1093/cid/ciae437. PMID 39180326

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from July 2019 to July 2023 at 56 sites in the US and Canada. Recruitment was performed by trained investigators and study coordinators.
Pre-assignment Details: A total of 793 participants were enrolled/signed informed consent of which 95 were screen failures.
  698 subjects were enrolled and were not screen failures. One participant was enrolled but not treated, therefore 697 participants received a dose of RBX2660.
Period: Overall Study
Arm/Group | Active
Started | 698
Completed | 635
Not Completed | 63

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- RBX2660: RBX2660 is a rectally administered microbiota suspension
  RBX2660: RBX2660 is a microbiota suspension administered rectally
Arm/Group | RBX2660
Number analyzed (Participants) | 697
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 359
  >=65 years | 338
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (17.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 487
  Male | 210
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 670
  Unknown or Not Reported | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 21
  White | 654
  More than one race | 4
  Unknown or Not Reported | 10
Region of Enrollment [Number; unit: participants]
  Canada | 117
  United States | 580

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of RBX2660 in Subjects With Recurrent CDI.
Description: Number of subjects with investigational product- and/or enema-related treatment-emergent adverse events (TEAEs).
Time Frame: Up to 6 months after last study treatment.
Population: Safety
Measure: Count of Participants; unit: Participants
Groups:
- Active Treatment: 1 enema of RBX2660
Arm/Group | Active Treatment
Number analyzed (Participants) | 697
Participants | 697

2. Secondary Outcome: Efficacy of RBX2660 Measured at 8 Weeks After Treatment.
Description: The absence of C. difficile diarrhea without the need for retreatment through 8 weeks after administration of the study treatment.
Time Frame: 8 weeks after completing the study treatment
Population: Modified Intent-to-Treat (MITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Active
Number analyzed (Participants) | 676
Participants | 499

3. Secondary Outcome: Sustained Clinical Response Through 6 Months After Treatment.
Description: Treatment success of the presenting CDI recurrence and no new CDI episodes for greater than 8 weeks through 6 months after completing a study treatment assessed by subject phone interview up to 6 months after the last study treatment.
Time Frame: 6 months after completing the study treatment
Population: Modified Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment
Number analyzed (Participants) | 499
Participants | 454

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Active
All-Cause Mortality (participants affected / at risk) | 6/697
Serious Adverse Events (participants affected / at risk) | 87/697
Other Adverse Events (participants affected / at risk) | 265/697
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=697)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2)
Cardiac failure (Cardiac disorders) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Spina bifida (Congenital, familial and genetic disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Upper gastrointestingal haemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Cardiac cirrhosis (Hepatobiliary disorders) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 21 (25)
Clostridium difficile colitis (Infections and infestations) | 6 (7)
Urosepsis (Infections and infestations) | 3 (3)
Diverticulitis (Infections and infestations) | 2 (2)
Clostridial sepsis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 2 (2)
Bacteraemia (Infections and infestations) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1)
Colonic abcess (Infections and infestations) | 1 (1)
Corona virus infection (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Infected bite (Infections and infestations) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 1 (1)
Osteomylitis (Infections and infestations) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 (1)
Streptococcal endocarditis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Post-tramatic pain (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Subarachnoid hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Alcoholic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrolvascular accident (Nervous system disorders) | 3 (3)
Encephalopathy (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (3)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1)
Alcoholism (Psychiatric disorders) | 1 (1)
Mental disorder (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 5 (5)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Colostomy (Surgical and medical procedures) | 1 (1)
Spinal nerve stimulator implantation (Surgical and medical procedures) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Shock (Vascular disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Ketosis (Metabolism and nutrition disorders) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Quadraparesis (Nervous system disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=697)
Diarrhoea (Gastrointestinal disorders) | 135 (172)
Abdominal pain (Gastrointestinal disorders) | 94 (116)
Nausea (Gastrointestinal disorders) | 61 (72)
Abdominal distension (Gastrointestinal disorders) | 45 (59)
Flatulence (Gastrointestinal disorders) | 39 (46)
Constipation (Gastrointestinal disorders) | 37 (46)
Urinary tract infection (Infections and infestations) | 41 (49)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT03931941/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/41/NCT03931941/SAP_001.pdf